CLINICAL TRIAL: NCT01167725
Title: Pilot / Phase III Randomized Trial Comparing Standard Systemic Therapy to Cytoreduction + Hyperthermic Intraperitoneal Mitomycin C + Standard Systemic Therapy in Patients With Limited Peritoneal Dissemination of Colon Adenocarcinoma
Brief Title: Standard Therapy With or Without Surgery and Mitomycin C in Treating Patients With Advanced Limited Peritoneal Dissemination of Colon Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000681540; WRAMC-8214, Z6091; CDR0000681540 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-01572 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer
Keywords: mucinous adenocarcinoma of the colon; stage III colon cancer; stage IV colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Bevacizumab; Cetuximab; Folfox protocol; Capecitabine; Fluorouracil; Irinotecan; Leucovorin; Mitomycin; Oxaliplatin

ARMS (2):
- Arm I (Active Comparator): Patients receive standard systemic therapy, at the discretion of patients' oncologist, comprising combinations of fluorouracil, leucovorin calcium, irinotecan hydrochloride, oxaliplatin, and/or capecitabine (including FOLFOX4, mFOLFOX6, CapeOx, or FOLFIRI), bevacizumab, or cetuximab. Treatment repeats in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may crossover to arm II.
  Interventions: Biological: bevacizumab; Biological: cetuximab; Drug: FOLFIRI regimen; Drug: FOLFOX regimen; Drug: capecitabine; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: oxaliplatin
- Arm II (Experimental): Patients undergo cytoreduction surgery and hyperthermic intraperitoneal mitomycin C over 45-90 minutes. Beginning 8 weeks after surgery, patients receive standard systemic therapy as in arm I. Treatment with systemic therapy repeats for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Biological: cetuximab; Drug: FOLFIRI regimen; Drug: FOLFOX regimen; Drug: capecitabine; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: mitomycin C; Drug: oxaliplatin; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Biological: bevacizumab — Given IV
Biological: cetuximab — Given IV
Drug: FOLFIRI regimen — Given IV
Drug: FOLFOX regimen — Given IV
Drug: capecitabine — Given IV
Drug: fluorouracil — Given IV
Drug: irinotecan hydrochloride — Given IV
Drug: leucovorin calcium — Given IV
Drug: mitomycin C — Given intraperitoneally
  Arms: Arm II
Drug: oxaliplatin — Given IV
Procedure: therapeutic conventional surgery — Patients undergo cytoreductive surgery
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Heating mitomycin C to several degrees above normal body temperature and infusing it into the area around the tumor may kill more tumor cells. Giving mitomycin C after surgery may kill any remaining tumor cells. It is not yet known whether standard therapy is more effective with or without surgery followed by mitomycin C.

PURPOSE: This randomized phase III trial is studying standard therapy with or without surgery and mitomycin C in treating patients with advanced limited peritoneal dissemination of colon cancer

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the overall survival (OS) of patients with advanced limited peritoneal dissemination of colon adenocarcinoma treated with systemic therapy with vs without cytoreduction surgery and hyperthermic intraperitoneal mitomycin C.
* To compare the relative OS at 1 year of patients treated with these regimens.

Secondary

* To compare the progression-free survival (PFS) of patients treated with these regimens.
* To compare the relative PFS at 1 year of patients treated with these regimens.
* To compare the quality of life of patients treated with these regimens.
* To compare the toxicity burden of these regimens in these patients.
* To compare the OS and PFS according to patients' peritoneal surface tumor genotype for the NAD(P)H (quinone oxidoreductase 1 [NQO1] 609C >T polymorphism [wild type vs heterozygous/homozygous mutant]) in patients treated with these regimens.
* To compare circulating tumor cells in patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to presentation (synchronous vs metachronous carcinomatosis), ECOG performance status (0 vs 1), disease volume (measurable vs non-measurable), prior first-line therapy for advanced disease (chemo-naïve vs prior first-line therapy), planned chemotherapy (oxaliplatin vs irinotecan vs fluorouracil/leucovorin calcium vs capecitabine), and planned biologic therapy (bevacizumab vs cetuximab vs none). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive standard systemic therapy, at the discretion of patients' oncologist, comprising combinations of fluorouracil, leucovorin calcium, irinotecan hydrochloride, oxaliplatin, and/or capecitabine (including FOLFOX4, mFOLFOX6, CapeOx, or FOLFIRI) with or without bevacizumab (beginning 4-6 weeks after major surgery) or cetuximab*. Treatment repeats in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may crossover to arm II.

NOTE: *For patients with KRAS wild-type tumors.

* Arm II: Patients undergo cytoreduction surgery and hyperthermic intraperitoneal mitomycin C over 45-90 minutes. Beginning 8 weeks after surgery, patients receive standard systemic therapy as in arm I. Treatment with systemic therapy repeats for 6 courses in the absence of disease progression or unacceptable toxicity.

Blood and tissue samples may be collected from patients for correlative studies.

Patients complete SF-36 Health Survey; Functional Assessment of Cancer Therapy-Colorectal (FACT-C); Feeling Sad, Down, or Depressed (CES-D); and a Brief Pain Inventory quality-of-life questionnaires at baseline and then periodically during study.

After completion of study therapy, patients are followed up periodically for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed colon adenocarcinoma meeting the following criteria:

  * Newly diagnosed disease
  * Advanced disease
  * Confirmed synchronous or metachronous limited peritoneal disease dissemination
  * No appendiceal or rectal cancer
  * No signet ring cell type
* Disease amenable to complete cytoreduction surgery as indicated by:

  * Peritoneal Cancer Index (PCI) ≤ 20 by helical CT scan and/or staging laparoscopy
  * No parenchymal hepatic metastases
  * No clinical (jaundice), biochemical (abnormally elevated serum bilirubin and/or alkaline phosphatase), or radiological (by ultrasound, CT scan, or MRI) biliary obstruction
  * No symptomatic malignant ascites requiring palliative paracentesis
  * Small volume of disease in the gastro-hepatic ligament defined by a < 5 cm mass in the epigastric region on cross-sectional imaging
  * No cross-sectional imaging findings indicative of multi-segmental (> 1 site) small bowel obstruction, small bowel loops matted together, or gross disease of the small bowel mesentery characterized by distortion, thickening, or loss of mesenteric vascular clarity
  * No clinical or radiological evidence of hematogenous or distant nodal (retroperitoneal, pelvic, mediastinal, peri-portal, or peri-aortic) metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* ANC > 1,200/mm³
* WBC > 4,000/mm³
* Platelet count 150,000/mm³
* INR ≤ 1.5

  * Patients on therapeutic anticoagulant for unrelated medical condition such as atrial fibrillation or anti-thrombocyte treatment allowed provided treatment can be withheld for operation
* Total serum bilirubin ≤ 1.5 mg/dL (> 1.5 mg/dL for patients with Gilbert syndrome)
* Alkaline phosphatase < 2.5 times upper limit of normal (ULN)
* AST < 1.5 times ULN
* Serum creatinine normal
* BUN normal
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No history of severe congestive heart failure or severe pulmonary disease

  * Patients who are status post-revascularization procedures with satisfactory cardiac function are eligible
* No acute myocardial infarction within the past 6 months
* No significant history of a medical problem or co-morbidity (e.g., severe congestive heart failure or active ischemic heart disease) that would preclude a major abdominal operation
* No concurrent second malignancy requiring systemic therapy
* No psychiatric or addictive disorders, or other conditions that would preclude the patient from meeting the study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior second-line systemic treatment for metastatic colon adenocarcinoma

  * Patients who received prior adjuvant therapy for colon adenocarcinoma and/or prior first-line systemic therapy for metastatic colon adenocarcinoma are eligible

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS)

SECONDARY OUTCOMES:
Progression-free survival (PFS)
Quality of life
Toxicity burden
Circulating tumor cells
Comparison of OS and PFS according to patients' peritoneal surface tumor genotype for the NAD(P)H

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Stojadinovic, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (2):
- United States (2):
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina